CLINICAL TRIAL: NCT02816385
Title: Study of Myocardial Contractility After Cardiac Surgery Under an Anterograde or Retrograde Cardioplegia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Pierre Wauthy, Head of clinic, Brugmann University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHUB-Retroplegie
Record Dates: First submitted 2016-04-20; First posted 2016-06-28 (Estimated); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Heart Arrest
Keywords: PV-loops (pressure-volume loops); Myocardial contractility; Cardioplegia; Induced
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antegrade Cardioplegia (Active Comparator): Coronary artery bypass grafting (CABG) surgery in patients with a normal left ventricular ejection fraction (FEVG)
  Interventions: Procedure: Antegrade cardioplegia
- Retrograde Cardioplegia (Experimental): Coronary artery bypass grafting (CABG) surgery in patients with a normal left ventricular ejection fraction (FEVG)
  Interventions: Procedure: Retrograde cardioplegia

INTERVENTIONS:
Procedure: Antegrade cardioplegia — Injection of the cardioplegia in the coronary arteries
  Arms: Antegrade Cardioplegia
Procedure: Retrograde cardioplegia — Injection of the cardioplegia in the venous system
  Arms: Retrograde Cardioplegia

SUMMARY:
Myocardial protection is a fundamental element for the safety of patients when performing cardiac surgery. For this purpose, cardioplegia were rapidly established in clinical practice to protect the myocardium when performing aortic clamp.

Cardioplegia are procedures to stop the contraction of myocardium. It is usually achieved with the use of chemicals ( cardioplegic solutions) or cold temperature (such as chilled perfusate). The composition of the cardioplegic solutions and their method of administration continuously changed over the years.

At the present date, cold blood cardioplegias are performed in the investigator's center. The investigators regularly use two modes of administration: either by an antegrade path (injection in the coronary arteries), or a retrograde one (injection in the venous system). At present, there are no elements supporting the superiority or inferiority of one path compared to another. The difficulty lies within a clear estimation of the contractility state of the ventricular cardiac muscle.

Technological developments in recent years provided a solution to this problem. The analysis of the pressure/volume curves generated by a ventricle allows an accurate quantification of the myocardial contractility. This requires the use of conductance catheters to accurately measure the ventricular volume and the ventricular pressure. The absolute ventricular contractility is then deduced with the help of a software.

The investigators intend to use this pressure-volume loops, obtained with conductance catheters, to compare the contractility of the right heart ventricle after antegrade vs retrograde cardioplegia.

ELIGIBILITY:
Inclusion Criteria:

* Need for myocardial revascularisation
* Normal FEVG ( > 50%)

Exclusion Criteria:

* Valvulopathy
* Associated procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Contractility index of the right ventricle | Baseline
  Cardiac surgery is performed according to the standard of care. The intraventricular pressure and the ventricular volume, measured with a conductance catheter, are combined within a software to compute the contractility index of the right ventricle. The baseline measure will be performed before the instauration of the extracorporeal blood circulation, during the cardiac surgery.
Contractility index of the right ventricle | immediately after discontinuation of the extracorporeal blood circulation (end of cardiac surgery according to standard of care - up to 4h)
  Cardiac surgery is performed according to the standard of care. The intraventricular pressure and the ventricular volume, measured with a conductance catheter, are combined within a software to compute the contractility index of the right ventricle. This will be measured at the end of the cardiac surgery, immediately after discontinuation of the extracorporeal circulation, with absence of inotropic support.
Contractility index of the right ventricle | 10 minutes after discontinuation of the extracorporeal blood circulation
  Cardiac surgery is performed according to the standard of care. The intraventricular pressure and the ventricular volume, measured with a conductance catheter, are combined within a software to compute the contractility index of the right ventricle. This will be measured at the end of the cardiac surgery, 10 minutes after discontinuation of the extracorporeal circulation, with absence of inotropic support.
Contractility index of the right ventricle | 20 minutes after discontinuation of the extracorporeal blood circulation
  Cardiac surgery is performed according to the standard of care. The intraventricular pressure and the ventricular volume, measured with a conductance catheter, are combined within a software to compute the contractility index of the right ventricle. This will be measured at the end of the cardiac surgery, 20 minutes after discontinuation of the extracorporeal circulation, with absence of inotropic support.

SECONDARY OUTCOMES:
Troponin post operative level | 6h post surgery
  The investigators would like to measure post operative troponin levels as a biological marker of myocardial protection
Troponin post operative level | 12h post surgery
  The investigators would like to measure post operative troponin as a biological marker of myocardial protection.
Troponin post operative level | 24h post surgery
  The investigators would like to measure post operative troponin as a biological marker of myocardial protection.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Wauthy, MD, Pr, Principal Investigator — CHU Brugmann; Alessandro Falchetti, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium